CLINICAL TRIAL: NCT06695624
Title: Investigation of the Effectiveness of Bilateral Endoscopic Sphenopalatine Ganglion Block in Management of Postoperative Pain After Septoplasty
Brief Title: Effectiveness of Bilateral Endoscopic Sphenopalatine Ganglion Block on Postoperative Pain After Septoplasty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Senay Goksu, specialist doctor, Umraniye Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SPGB-FULYA
Record Dates: First submitted 2024-11-12; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Pain
Keywords: sphenopalatine ganglion block; septoplasty; postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Sphenopalatine Ganglion Block

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group with sphenopalatine ganglion block (Active Comparator): Sphenopalatine ganglion block will be performed for participants undergoing septoplasty.
  Interventions: Procedure: Sphenopalatine Ganglion Block
- group without sphenopalatine ganglion block (No Intervention): Sphenopalatine ganglion block will not be performed for participants undergoing septoplasty

INTERVENTIONS:
Procedure: Sphenopalatine Ganglion Block — Sphenopalatine ganglion block group 4cc (80mg) 2% lidocaine + 1cc (4mg) dexamethasone in total 5cc volume will be prepared under sterile conditions before the procedure, 2.5 cc will be given to both nostrils. Sphenopalatine ganglion block will be applied by transnasal endoscopic method.
  Arms: group with sphenopalatine ganglion block

SUMMARY:
The aim of this clinical study will investigate the efficacy of sphenopalatine ganglion block in the treatment of postoperative pain.it will also be learnt whether it reduces the consumption of analgesics in postoperative pain.The main questions it aims to answer are:

Will the participants' need for painkillers decrease after the operation? Can sphenopalatine ganglion block be used for postoperative pain after septoplasty? The researchers will compare 2 groups with and without sphenopalatine ganglion block to see the effectiveness of sphenopalatine ganglion block.

Participants will:

Read the information Participants have been given about the sphenopalatine ganglion block.

In case of any side effects, please contact participant's doctor.

DETAILED DESCRIPTION:
This randomised controlled study will be conducted in Umraniye Training and Research Hospital operating room between November 2024 and January 2025 after obtaining ethics committee and patient consent. Each patient will be informed about the procedures to be performed during anaesthesia and surgery and signed informed consent will be obtained before the procedure. Patients will undergo septoplasty by the same otolaryngology team.

A total of 50 participants (25 envelopes each with Group 1 and Group 2 written inside) will be kept closed for the patients participating in the study. Upon the patient's fulfilment of the conditions suitable for the study, it will be randomly determined which group he/she will be included in. Thanks to this randomisation, conscious or unconscious manipulations in the selection of patients to the study group will be prevented.

ELIGIBILITY:
Inclusion Criteria:

* Participants who will undergo septoplasty
* 18 to 50 years old
* ASA score 1 or 2

Exclusion Criteria:

* Under 18 or over 50 years of age
* ASA score III and above patient group
* The patient is allergic to any of the drugs used
* The patient has a contraindication to any of the drugs used
* Use of anticoagulant medication
* Failure of the patient to give consent
* Being pregnant
* Those with GCS retardation such as dementia, mental retardation
* Those with diagnosed headache

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale | 24 hours
  Zero is equivalent to no pain and 10 indicates the worst possible pain.
total amount of tramadol consumption | 24 hours
  Total tramadol consumption will be recorded in the postoperative period by fitting participants with a patient-controlled analgesia device.

CONTACTS AND LOCATIONS:
Overall Officials: şenay göksu, MD, Principal Investigator — Umraniye Education and Research Hospital Collaborators:

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Qudah M. Endoscopic sphenopalatine ganglion blockade efficacy in pain control after endoscopic sinus surgery. Int Forum Allergy Rhinol. 2016 Mar;6(3):334-8. doi: 10.1002/alr.21644. Epub 2015 Sep 15. PMID 26370724
- [Background] Ekici NY, Alagoz S. The effectiveness of endoscopic sphenopalatine ganglion block in management of postoperative pain after septal surgery. Int Forum Allergy Rhinol. 2019 Dec;9(12):1521-1525. doi: 10.1002/alr.22411. Epub 2019 Sep 5. PMID 31487422